CLINICAL TRIAL: NCT00243152
Title: Evaluation of Lamotrigine on Neuropathic Facial Pain Using fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain and Analgesia Imaging and Neuroscience Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, David Borsook, M.D., Ph.D., Dr., Pain and Analgesia Imaging and Neuroscience Group
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Facial Neuropathy/lamotrigine
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Facial Neuropathy
Keywords: pain; neuropathic; face; trigeminal
MeSH Terms: conditions — Facial Nerve Diseases; Pain; Facies | interventions — Lamotrigine; lipoarabinomannan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine to Placebo Crossover (Active Comparator): The drug lamotrigine will be given for 9 weeks prior to imaging session 1. A rescue drug, Gabapentin, will be provided for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. After a taper and washout, placebo (cross over) will be administered. At the end of the trial (after imaging session 2), a taper for placebo will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Interventions: Drug: Lamotrigine
- Placebo to Lamotrigine Crossover (Active Comparator): The placebo will be given for 9 weeks prior to imaging session 1. A rescue drug, Gabapentin, will be provided for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. After a taper and washout, the drug lamotrigine (cross over) will be administered. At the end of the trial (after imaging session 2), a taper for drug will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Interventions: Drug: Placebo (for Lamotrigine)

INTERVENTIONS:
Drug: Lamotrigine — : 25mg and 50mg tablets
  Other Names: LAMO; LAM
  Arms: Lamotrigine to Placebo Crossover
Drug: Placebo (for Lamotrigine) — Sugar pill manufactured to mimic Lamotrigine tablets
  Other Names: Placebo
  Arms: Placebo to Lamotrigine Crossover

SUMMARY:
The aim of this project is to evaluate the effects of the anticonvulsant drug lamotrigine (trade name Lamictal) on neuropathic facial pain or neuralgia using functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
Currently there are no pharmacological agents that can control neuropathic pain akin to the efficacy of antibiotics for bacterial infection. All current neuropathic pain drugs have approximately the same efficacy of less than 30% in controlled trials, and many of these drugs do not have known mechanisms of action. fMRI studies may provide insight into how brain circuitry is altered by chronic pain, and how these drugs act on altered circuitry. The trigeminal system in particular offers unique advantages for studying such alterations, including a large central representation and high degree of somatotopy. The administration of lamotrigine to neuropathic pain patients in conjunction with fMRI will allow us to compare subjective ratings of pain with objective measures of neural activity during increased conditions of allodynia/hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Right-handed non-smokers
* Diagnosed with facial pain
* Continuous pain for more than 3 months
* Spontaneous pain greater than 3 of 10
* Allodynia to brush greater than 5 of 10

Exclusion Criteria:

* Medications
* Depression
* Significant medical problems
* Claustrophobia
* Abnormal EKG
* Significant drug or alcohol history
* Positive drug screen
* Weight greater than 285 lbs
* History of allergy to anticonvulsants
* Tattoos with metallic ink on upper body
* Any neurostimulator devices, or metal cochlear, ocular, or cardiac implants or other metal near vital areas
* Exposure to shrapnel or metal filings
* Other metallic surgical hardware

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2005-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Borsook, M.D., Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital Neuroimaging Center, 115 Mill Street, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Becerra L, Breiter HC, Wise R, Gonzalez RG, Borsook D. Reward circuitry activation by noxious thermal stimuli. Neuron. 2001 Dec 6;32(5):927-46. doi: 10.1016/s0896-6273(01)00533-5. PMID 11738036
- [Background] Zakrzewska JM, Chaudhry Z, Nurmikko TJ, Patton DW, Mullens LE. Lamotrigine (lamictal) in refractory trigeminal neuralgia: results from a double-blind placebo controlled crossover trial. Pain. 1997 Nov;73(2):223-230. doi: 10.1016/S0304-3959(97)00104-8. PMID 9415509
- [Background] Petersen KL, Maloney A, Hoke F, Dahl JB, Rowbotham MC. A randomized study of the effect of oral lamotrigine and hydromorphone on pain and hyperalgesia following heat/capsaicin sensitization. J Pain. 2003 Sep;4(7):400-6. doi: 10.1016/s1526-5900(03)00718-1. PMID 14622682
- [Result] Scrivani S, Wallin D, Moulton EA, Cole S, Wasan AD, Lockerman L, Bajwa Z, Upadhyay J, Becerra L, Borsook D. A fMRI evaluation of lamotrigine for the treatment of trigeminal neuropathic pain: pilot study. Pain Med. 2010 Jun;11(6):920-41. doi: 10.1111/j.1526-4637.2010.00859.x. Epub 2010 May 11. PMID 20492571
- See also: P.A.I.N. Group article — https://painandthebrain.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited adult males and females ages 18 to 60 with diagnosed facial neuropathic pain.
Groups:
- Lamotrigine to Placebo Crossover: The drug lamotrigine taken 9 weeks prior to imaging session 1. A rescue drug, Gabapentin, provided during both arms of the study for pain control. Patients taper off the Gabapentin 2 weeks before each scan date. After a taper and washout period placebo (cross over) will be administered. At the end of the trial (after imaging session 2), a taper for placebo will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Lamotrigine: : 25mg and 50mg tablets
- Placebo to Lamotrigine Crossover: Placebo is taken 9 weeks prior to imaging session 1. A rescue drug, Gabapentin, provided during both arms of the study for pain control. Patients taper off the Gabapentin 2 weeks before each scan date. After a taper and washout period the drug, Lamotrigine (cross over), will be administered. At the end of the trial (after imaging session 2), a taper for drug will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
Period: Overall Study
Arm/Group | Lamotrigine to Placebo Crossover | Placebo to Lamotrigine Crossover
Started | 3 | 3
Scan 1: Drug or Placebo | 3 | 3
Scan 2: Placebo or Drug | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Both male and female adults ages 18 to 60 years old who are right-handed and non-smokers. Participants must be diagnosed with facial pain that has been continuous for more than 3 months. Their spontaneous pain must be great than 3 of 10 and their allodynia to brush must be greater than 5 of 10.
Groups:
- Lamotrigine: The drug lamotrigine or placebo will be given for 9 weeks prior to imaging session 1. A rescue drug, Gabapentin, will be provided during both arms of the study for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. After a taper and washout period lamotrigine or placebo (cross over) will be administered. At the end of the trial (after imaging session 2), a taper for drug/placebo will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Lamotrigine: : 25mg and 50mg tablets
Arm/Group | Lamotrigine
Number analyzed (Participants) | 6
Age, Customized [Number; unit: participants]
  Ages 18 to 60 Years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6
Diagnosed with facial pain [Number; unit: participants] | 6
Continuous pain for more than 3 months [Number; unit: participants] | 6
Spontaneous pain greater than 3 of 10 [Number; unit: participants] — Pain Scale Description: 0-10 rating scale where 0 indicates no pain and 10 indicates the highest pain
  participants | 6
Allodynia brush greater than 5 of 10 [Number; unit: participants] — Pain Scale Description: 0-10 rating scale where 0 indicates no pain and 10 indicates the highest pain
  participants | 6
Right-handed [Number; unit: participants] | 6
Non-smokers [Number; unit: participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygenation Level-dependent (BOLD) Changes in Neural Pain Circuitry Following Treatment With Lamotrigine During Experimentally Induced Pain States
Description: fMRI scans acquired Stimuli Type: Brush Stimulation Regions: Face (V2) Right and Left Sides Rating: Pain/ unpleasantness fMRI scans acquired Stimuli Type: Cold, threshold -1°C Stimulation Regions: Face (V2) Right and Left Sides Rating: Pain/ unpleasantness **Extra time allotted for probe repositioning** fMRI scans acquired Stimuli Type: Heat, threshold +1°C Stimulation Regions: Face (V2) Right and Left Sides Rating: Pain/ unpleasantness **Extra time allotted for probe repositioning** Cortical, subcortical, and brain stem sensory regions Z-scores Increase or decrease in activation as affected by the drug
Time Frame: Week 10 during scanning session
Population: The data's primary comparisons no longer exists per intervention.
Measure: Number; unit: Z-statistic
Groups:
- Lamotrigine vs Placebo: The drug lamotrigine will be given for 9 weeks prior to imaging session. A rescue drug, Gabapentin, will be provided for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. Placebo will be administered in another imaging session. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
Arm/Group | Lamotrigine vs Placebo
Number analyzed (Participants) | 6
Z-statistic
  Heat Affected Thalamus (10,-14,8) | -2.9294
  Heat Affected Post-Central (-56,-12,28) | -2.7323
  Cold Affected Post-Central (68, -8, 32) | -2.5114
  Cold Affected Thalamus (-4, -8, 0) | -3.033
  Brush Affected Post-Central (66,-16,14) | 3.905
  Brush Affected Thalamus (-14,-22, 4) | -3.791
  Brush Affected Spinal Trigeminal Nucles(2,-48,-68) | 2.9058

2. Secondary Outcome: Subjective Ratings of Pain During Magnetic Resonance Scanning
Description: Quantitative Sensory Testing (QST)
  Stimuli Type: Heat, Cold, Brush Stimulation Regions: Face Affected and contralateral Unaffected mirror area Rating: Pain/ unpleasantness Stimuli Type: Cold, threshold -1°C Stimulation Regions: Face Affected and contralateral Unaffected mirror area Rating: Pain/ unpleasantness Stimuli Type: Heat, threshold +1°C Stimulation Regions: Face Affected and contralateral Unaffected mirror area Rating: Pain/ unpleasantness
  Ratings on a likert scale of 0-10 with 0 being defined as no pain and 10 being defined as worst possible pain
Time Frame: week 10 (during the scan)
Measure: Mean (Standard Deviation); unit: scores on a pain scale
Groups:
- Placebo: The placebo will be given for 9 weeks prior to imaging session. A rescue drug, Gabapentin, will be provided for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. At the end of the trial (after imaging session 2), a taper for drug will be given. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Placebo (for Lamotrigine): Sugar pill manufactured to mimic Lamotrigine tablets
- Lamotrigine: The drug lamotrigine will be given for 9 weeks prior to imaging session. A rescue drug, Gabapentin, will be provided for pain control. Patients will taper off the Gabapentin 2 weeks before each scan date. Patients will be required to maintain a pain diary during the study, documenting the perceived effects of the drug on the severity of their pain and keeping track of their subjective pain ratings day to day. Patients will also complete the McGill Pain Questionnaire at each visit.
  Lamotrigine: : 25mg and 50mg tablets
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 6 | 6
scores on a pain scale
  Heat Affected | 5.5 (2) | 3.2 (1.5)
  Heat Unaffected | 4 (3) | 3 (2)
  Cold Affected | 2.5 (1.2) | 2.1 (1.5)
  Cold Unaffected | 1.1 (1) | 2.2 (1.75)
  Brush Affected | 3.9 (2.1) | 2.8 (2.8)
  Brush Unaffected | .4 (.3) | 1.2 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine; Visual analog scale (VAS) ratings in the scanner. Measures of pain ratings to evoked stimuli during scanning for heat applied to the affected side; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Lamotrigine; VAS rating in the scanner. Measures of pain rating to evoke stimuli during scanning for heat applied to the unaffected side; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs Lamotrigine; VAS rating in the scanner. Measures of pain rating to evoke stimuli during scanning for cold applied to the affected side; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs Lamotrigine; VAS rating in the scanner. Measures of pain rating to evoke stimuli during scanning for cold applied to the unaffected side; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs Lamotrigine; VAS rating in the scanner. Measures of pain rating to evoke stimuli during scanning for brush applied to the affected side; Test type: Superiority; p > 0.05, t-test, 2 sided
Statistical Analysis 6: Comparison: Placebo vs Lamotrigine; VAS rating in the scanner. Measures of pain rating to evoke stimuli during scanning for brush applied to the unaffected side; Test type: Superiority; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Lamotrigine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Every effort was made to obtain the data presented in outcome measure 2. However only the data in the publication is available, estimates were made based on the figures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No